CLINICAL TRIAL: NCT04214886
Title: Dose Escalation Study of CD19 Chimeric Antigen Receptor (CAR) T Cells With a CD34 Selection Marker in Adults With Recurrent or Refractory B Cell Malignancies
Brief Title: CD19 Chimeric Antigen Receptor (CAR) T Cells for Adults With Recurrent or Refractory B Cell Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Leukemia Research Foundation (Unknown)
Responsible Party: Principal Investigator, Nasheed Hossain, MD, Assistant Professor, Loyola University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 212594
Record Dates: First submitted 2019-12-16; First posted 2020-01-02 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: B-Cell Acute Lymphoblastic Leukemia, Adult; B-cell Lymphoma Refractory; B-cell Lymphoma Recurrent
Keywords: Leukemia; Lymphoma; CAR T; Chimeric; CD19
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia; Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Autologous peripheral blood mononuclear cell (PBMC) will be obtained by leukapheresis over one day. Daily intravenous (IV) infusion of fludarabine and cyclophosphamide for total of 3 days (Days -5, -4, -3). The dose of cyclophosphamide will be given at 500mg/m2. The dose of fludarabine will be given at 30mg/m2. CD19-CD34 CAR transduced T cells administration will follow a Phase I dose escalation design. Each Cohort will start will with the goal of accruing three participants to determine the dose limiting toxicities. Once the maximum tolerated dose is established, an expansion cohort will be treated to include a total of 6 participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CAR 5 x 105 transduced T cells/kg (Dose Level -1) (Experimental): Autologous peripheral blood mononuclear cell (PBMC) will be obtained by leukapheresis over one day. Daily intravenous (IV) infusion of fludarabine and cyclophosphamide for total of 3 days (Days -5, -4, -3). The dose of cyclophosphamide will be given at 500mg/m2. The dose of fludarabine will be given at 30mg/m2. CD19-CD34 CAR transduced T cells will be administered IV at a dose level of 5 x 105 transduced T cells/kg.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD19-CD34 CAR transduced T cells
- CAR 1 x 106 transduced T cells/kg (Dose Level 1) (Experimental): Autologous peripheral blood mononuclear cell (PBMC) will be obtained by leukapheresis over one day. Daily intravenous (IV) infusion of fludarabine and cyclophosphamide for total of 3 days (Days -5, -4, -3). The dose of cyclophosphamide will be given at 500mg/m2. The dose of fludarabine will be given at 30mg/m2. CD19-CD34 CAR transduced T cells will be administered IV at a dose level of 1 x 106 transduced T cells/kg.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD19-CD34 CAR transduced T cells
- CAR 1.5 x 106 transduced T cells/kg (Dose Level 2) (Experimental): Autologous peripheral blood mononuclear cell (PBMC) will be obtained by leukapheresis over one day. Daily intravenous (IV) infusion of fludarabine and cyclophosphamide for total of 3 days (Days -5, -4, -3). The dose of cyclophosphamide will be given at 500mg/m2. The dose of fludarabine will be given at 30mg/m2. CD19-CD34 CAR transduced T cells will be administered IV at a dose level of 1.5 x 106 transduced T cells/kg.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD19-CD34 CAR transduced T cells
- CAR 2 x 106 transduced T cells/kg (Dose Level 3) (Experimental): Autologous peripheral blood mononuclear cell (PBMC) will be obtained by leukapheresis over one day. Daily intravenous (IV) infusion of fludarabine and cyclophosphamide for total of 3 days (Days -5, -4, -3). The dose of cyclophosphamide will be given at 500mg/m2. The dose of fludarabine will be given at 30mg/m2. CD19-CD34 CAR transduced T cells will be administered IV at a dose level of 2 x 106 transduced T cells/kg.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CD19-CD34 CAR transduced T cells

INTERVENTIONS:
Drug: Fludarabine — Fludarabine is an anti-cancer drug acting as an antimetabolite that is used to treat leukemia and lymphoma cancers.
Drug: Cyclophosphamide — Cyclophosphamide is is an anti-cancer drug acting as an alkylating agent that is used to treat leukemia and lymphoma cancers.
Biological: CD19-CD34 CAR transduced T cells — CD19-CD34 CAR transduced T cells are the subject's own immune cells that target B cell markers on cancer cells.

SUMMARY:
In this protocol, the investigators hypothesize that modifying the process of producing CAR+ T-cells can help to improve responses and reduce toxicities. Building on previous in vitro studies that have shown successful production of CAR+ T-cells using a new production approach, the investigators are now studying the ability to produce these CAR+ T-cells and determine how well they work in the clinical setting.

DETAILED DESCRIPTION:
Autologous peripheral blood mononuclear cell (PBMC) will be obtained by leukapheresis over one day and the cells will be transduced with an in house designed CAR retroviral vector. Participants will receive daily intravenous (IV) infusion of lymphodepleting regimen of fludarabine and cyclophosphamide for total of 3 days (Days -5, -4, -3). The dose of cyclophosphamide will be given at 500mg/m2. The dose of fludarabine will be given at 30mg/m2. Participants will receive the CAR transduced T cells IV infusion in the BMT Inpatient Unit and remain admitted for close monitoring for at least the first 7 days following the cell infusion (D0 to Day +7), possibly longer if any side effects are encountered. The CAR transduced T cells will be escalated from 1 x 106 transduced T cells/kg (± 20%) to 2 x 106 transduced T cells/kg (± 20%) in a Phase I design, based on toxicity. Once discharged from the inpatient unit, for the next 7 days (Day +8 to Day +14) the patients will be evaluated in the High Dose Unit (labs and physical exam) to screen for toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than or equal to 18 years of age.
* Participants must have Eastern cooperative oncology group (ECOG) performance status of 0 or 1, or Karnofsky greater than or equal to 80%
* Participants must have been diagnosed with histologically confirmed aggressive B cell NHL that is refractory / recurrent.
* Participants must have been diagnosed with histologically confirmed B-ALL that is refractory / recurrent.
* All subjects must have evaluable or measurable disease; subjects with lymphoma must have evaluable or measurable disease according to the revised IWG Response Criteria for Malignant Lymphoma. Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy. ALL patients must have at least 5% blasts in the bone marrow
* Adequate performance status; adequate organ and marrow function as defined by (supportive care is allowed per institutional standards, i.e. filgrastim, transfusion):
* ANC ≥ 750/uL*
* Platelet count ≥ 50,000/uL*
* Absolute lymphocyte count ≥ 150/uL*
* Adequate renal, hepatic, pulmonary and cardiac function defined as:

  * SaO2 ≥ 92% on room air
  * Creatinine ≤ 2 mg/dL or Creatinine Clearance ≥ 60 mL/min (as estimated by Cockcroft Gault)
  * Total bilirubin ≤ 1.5 mg/dL (except in subjects with Gilbert's disease) (Elevations related to leukemia or lymphoma involvement of the liver will not disqualify a subject)
  * Serum ALT/AST ≤3x ULN or ≤5X if there is hepatic involvement due to malignancy
  * Cardiac ejection fraction (LVEF) ≥ 45%)
* Subjects with ALL or B-NHL with CNS1, or CNS1a, 2b, 2c are eligible only in the absence of neurologic symptoms suggestive of CNS disease involvement such as cranial nerve palsy.
* If patients previously had CNS disease and are disease free after treatment with no clinical concerns for recurrent disease they are eligible for enrollment.
* Subjects with history of allogeneic SCT must be at least 100 days from SCT, have no evidence of Graft versus Host Disease (GvHD), and no longer taking immunosuppressive agents for at least 30 days prior to enrollment. However, patients with grade 1 skin GVHD or low grade cGHVD <3 who are not requiring systemic therapy are eligible.
* Females of child bearing potential and males of child fathering potential must be willing to practice birth control during and for 4 months post therapy.
* Females of child bearing potential must have negative pregnancy test.
* Must meet wash out period since prior therapies.

  * At least 2 weeks or 5 half-lives, whichever is shorter, must have elapsed since any prior systemic therapy at the time the subject is planned for leukapheresis, except for systemic inhibitory/stimulatory immune checkpoint therapy, which requires 5 half-lives
* Must have recovered from acute side effects from prior therapy to meet eligibility.
* If had prior CAR therapy, 30 days must have elapsed prior to apheresis; may not have evidence of persistence of CAR T cells in blood samples (circulating levels of genetically modified cells of ≥ 5% by flow cytometry)
* No active HIV or active HBV/HCV infection. Patients with history of HBV or HCV who are PCR negative after appropriate therapy are eligible. Patients may not have any other uncontrolled, symptomatic, intercurrent illness.
* No history of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study.
* No active CNS disorder, or history of MI, cardiac angioplasty or stenting, unstable angina or other clinically significant cardiac disease with 12 months of enrollment, or have cardiac atrial or ventricular lymphoma involvement.
* Not receiving anticoagulation therapy
* Not have primary immunodeficiency or history of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years

Exclusion Criteria:

* Participants must not have an active bacterial, viral, fungal or other infection.
* Participants must not have a history of HIV or current hepatitis B or hepatitis C virus
* Participants must not have a history of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment, or have cardiac atrial or cardiac ventricular lymphoma involvement.
* No history of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study.
* No active CNS disorder, or history of MI, cardiac angioplasty or stenting, unstable angina or other clinically significant cardiac disease with 12 months of enrollment, or have cardiac atrial or ventricular lymphoma involvement.
* Not receiving anticoagulation therapy
* Not have primary immunodeficiency or history of autoimmune disease (e.g. Crohns, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years
* History of malignancy other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, and breast) unless disease free for at least 1 year. Patients who are on adjuvant therapy with no evidence of active disease are deemed eligible for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful production of CD19-CD34 CAR product that meet predefined release criteria (cell viability/cell number/transduction efficiency/negative sterility and viral testing) for enrolled patients | 18 months
  24 participants evaluated for determination of the feasibility of producing CD19-CD34 CAR T cells meeting the established release criteria
Adverse events | 15 years
  24 participants evaluated for adverse event and grading by using CTCAE v.5.0 to determine the maximal tolerated dose of CD19-CD34 CAR T cells with chemotherapy conditioning regimen for patients that have recurrent or refractory B cell malignancies

SECONDARY OUTCOMES:
Response to treatment | 24 months
  24 participants evaluated for response to treatment by testing using PET/CT for lymphoma and using bone marrow aspirate for leukemia.
Progression free survival | 24 months
  24 participants evaluated for progression by testing using PET/CT for lymphoma and using bone marrow aspirate for leukemia.
Overall survival | 15 years
  24 participants evaluated for overall survival by clinical visit

OTHER OUTCOMES:
Immune response | 15 years
  24 participants evaluated for immune response by blood tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nasheed Hossain, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No